CLINICAL TRIAL: NCT06491953
Title: Impact of SGLT2-inhibitors on Post Contrast Acute Kidney Injury in Acute Coronary Syndrome Patients Receiving Invasive Strategy
Brief Title: SGLT2-inhibitors on PC-AKI
Status: Active, not recruiting | Type: Observational
Sponsor: Shenyang Northern Hospital (Other)
Responsible Party: Principal Investigator, Han Yaling, Prof., Shenyang Northern Hospital
Other Study IDs: TIMING-AKI V1.0
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Impact of SGLT2-inhibitors on PC-AKI in ACS Patients Receiving Invasive Strategy
MeSH Terms: interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients receiving invasive treatment: Patients receiving PCI or CAG were enrolled to evaluate the impact of SGLT-2 inhibitors use or not use and duration of SGLT-2 inhibitors administration
  Interventions: Drug: SGLT-2 inhibitors

INTERVENTIONS:
Drug: SGLT-2 inhibitors — SGLT-2 inhibitors use or not use； the duration of SGLT-2 inhibitors use

SUMMARY:
Percutaneous coronary intervention (PCI) is one of the most common invasive strategies employed in the diagnosis and treatment of coronary artery disease (CAD) patients. Invasive procedures necessitate the use of iodine-based contrast agents, which could lead to post contrast acute kidney injury (PC-AKI).

Sodium-glucose cotransporter 2 (SGLT-2) inhibitors, as a class of oral antidiabetic medications, function by inhibiting SGLT-2, preventing the reabsorption of filtered glucose by the kidneys and thereby increasing glucose excretion in urine. In recent years, a series of studies including EMPA-REG OUTCOME, CREDENCE, DAPA-CKD, DECLARE-TIMI 58, and the CANVAS program have consistently demonstrated that SGLT-2 inhibitors not only effectively improve renal function and slow the progression of chronic kidney disease (CKD), but also significantly reduce the risk of cardiovascular adverse events. Nevertheless, due to their osmotic diuretic effect, SGLT-2 inhibitors can lead to a reduction in renal blood volume within the early phase of application (within two weeks), temporarily augmenting the renal workload and resulting in a decrease in estimated glomerular filtration rate (eGFR).

Consequently, there remains a need to ascertain the specific role of SGLT-2 inhibitors in the prevention of PC-AKI and provide evidence-based support for their application in this context.

ELIGIBILITY:
Inclusion Criteria:

* ACS patients undergoing invasive treatment (PCI or CAG)
* 18 ~ 80 years old adult patients
* Written informed consent provided

Exclusion Criteria:

* Administration of any iodinated CM within 14 days before CAG or PCI
* Hepatic dysfunction (ALT 3 times greater than upper normal limit)
* Thyreoid insufficiency
* Renal artery Stenosis (unilateral >70％ or bilateral stenosis>50％)
* Known allergy to any of the study drugs or devices (iodinated CM, etc.)
* Pregnancy or lactation
* Contraindications for the use of SGLT-2 inhibitors, such as severe renal insufficiency (eGFR <30 mL/min/1.73m2 or currently on dialysis), type 1 diabetes mellitus, severe infection, etc.)
* Any condition which might interfere with study compliance, or otherwise unsuitable for study participation as judged by the investigators

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ACS patients aged 18-80 years old receiving invasive treatment were enrolled.
Sampling Method: Probability Sample
Enrollment: 3600 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2026-05-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of Post contrast acute kidney injury (PC-AKI) | 48 hours after procedure
  PC-AKI was defined by the European Society of Genitourinary Radiology (EUSR): increase in serum creatinine by ≥ 0.3 mg/dl (≥ 26.5 μmol/l) within 48 hours or increase in serum creatinine (SCr) to ≥ 1.5 times the known baseline

SECONDARY OUTCOMES:
Major adverse cardiovascular and cerebrovascular events(MACCE) | up to 12 months
  Cardiovascular death, non-fatal myocardial infarction, stroke, or ischemic-driven target vessel revascularization
All-cause mortality | up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Northern Theater Command, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No